CLINICAL TRIAL: NCT02426801
Title: Feasibility of a Mobile Intervention to Increase Adherence to Asthma Medication Among Children Age 11 to 19 in an Urban Setting
Brief Title: Feasibility Trial of a Mobile Adherence Tool for Adolescents With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CoheroHealth (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014_Spring_Feasibility
Record Dates: First submitted 2015-04-07; First posted 2015-04-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: Patient Compliance; Mobile Applications; Medication Adherence
MeSH Terms: conditions — Asthma; Patient Compliance; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Patients in this arm were given no intervention. Their self-reported medication adherence was assessed at the baseline (week 0) and follow-up (week 12) visits but during the study period they did not receive any intervention.
- Medication Sensor Only (Sham Comparator): These patients received the medication use sensor (sham intervention) and downloaded a sham version of the mobile app. Thus, the medication use from these patients was able to be recorded but the patients did not receive reminders or incentives or the ability to see their medication use via the real mobile app.
  Intervention: inhaler sensor
  Interventions: Device: Inhaler sensor
- Medication Sensor and Mobile App (Experimental): These patients received the medication use sensor and the mobile app with reminders (intervention arm).
  Interventions: inhaler sensor and mobile application for asthma adherence
  Interventions: Device: Inhaler sensor; Behavioral: Mobile application for asthma adherence

INTERVENTIONS:
Device: Inhaler sensor — Inhaler sensor strap that tracks inhaler use via a pressure sensitive switch.
  Arms: Medication Sensor Only; Medication Sensor and Mobile App
Behavioral: Mobile application for asthma adherence — Mobile phone application that sends reminders, allows patients to see their medication use, and provides points and other incentives for medication use.
  Arms: Medication Sensor and Mobile App

SUMMARY:
The purpose of this study is to assess the feasibility of using a mobile health intervention to improve adherence to asthma medication among adolescents in an urban clinic setting. The intervention consists of an inhaler sensor strap to monitor asthma inhaler use and a mobile phone application to remind and incentivize patients to use their medication. This study will assess the feasibility and acceptability of this intervention to patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-19
* Asthma diagnosis
* Currently on a daily controller medication for Asthma
* English-speaking

Exclusion Criteria:

* Pregnant
* Foster Care
* Emancipated minor

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Evidence of ability to monitor medication use at home via a sensor strap | 12 weeks
  Ability to measure medication use via the sensor strap and upload that information to the HIPAA (Health Insurance Portability and Accountability Act) compliant server.

SECONDARY OUTCOMES:
Patient feedback for improved design of a mobile adherence tool | 12 weeks
  Feedback from patients on the design of the inhaler sensor and mobile app including aesthetics and ease of use.
Acceptability of mobile adherence strategy for adolescents with asthma (Based on questions as part of baseline/followup visits and focus group.) | 12 weeks
  Based on questions as part of baseline/followup visits and focus group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Parides, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Andrew M Ting, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

REFERENCES:
- [Background] Stern L, Berman J, Lumry W, Katz L, Wang L, Rosenblatt L, Doyle JJ. Medication compliance and disease exacerbation in patients with asthma: a retrospective study of managed care data. Ann Allergy Asthma Immunol. 2006 Sep;97(3):402-8. doi: 10.1016/S1081-1206(10)60808-3. PMID 17042149
- [Background] Claxton AJ, Cramer J, Pierce C. A systematic review of the associations between dose regimens and medication compliance. Clin Ther. 2001 Aug;23(8):1296-310. doi: 10.1016/s0149-2918(01)80109-0. PMID 11558866
- [Background] Chapman KR, Walker L, Cluley S, Fabbri L. Improving patient compliance with asthma therapy. Respir Med. 2000 Jan;94(1):2-9. doi: 10.1053/rmed.1999.0667. PMID 10714473
- [Background] Einarson TR. Drug-related hospital admissions. Ann Pharmacother. 1993 Jul-Aug;27(7-8):832-40. doi: 10.1177/106002809302700702. PMID 8364259
- [Background] Bender BG, Rand C. Medication non-adherence and asthma treatment cost. Curr Opin Allergy Clin Immunol. 2004 Jun;4(3):191-5. doi: 10.1097/00130832-200406000-00009. PMID 15126940
- [Background] Lasmar L, Camargos P, Champs NS, Fonseca MT, Fontes MJ, Ibiapina C, Alvim C, Moura JA. Adherence rate to inhaled corticosteroids and their impact on asthma control. Allergy. 2009 May;64(5):784-9. doi: 10.1111/j.1398-9995.2008.01877.x. Epub 2009 Jan 21. PMID 19183166
- [Background] Patrick H, Williams GC. Self-determination theory: its application to health behavior and complementarity with motivational interviewing. Int J Behav Nutr Phys Act. 2012 Mar 2;9:18. doi: 10.1186/1479-5868-9-18. PMID 22385676
- [Background] McCallum S. Gamification and serious games for personalized health. Stud Health Technol Inform. 2012;177:85-96. PMID 22942036
- [Background] Csikszentmihalyi M, Rathunde K. The measurement of flow in everyday life: toward a theory of emergent motivation. Nebr Symp Motiv. 1992;40:57-97. No abstract available. PMID 1340523